CLINICAL TRIAL: NCT02151331
Title: Improving Mental Health Outcomes: Building an Adaptive Implementation
Brief Title: Improving Mental Health Outcomes: Building an Adaptive Implementation Strategy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor requested termination due to low recruitment numbers
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy M. Kilbourne, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01MH099898-01A1 (NIH); 1R01MH099898-01A1 (NIH)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-11

CONDITIONS: Bipolar Disorder; Depression; Mood Disorder
Keywords: Chronic care model; Mood disorders; Adaptive implementation
MeSH Terms: conditions — Bipolar Disorder; Depression; Mood Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- REP + EF (Experimental): Replication Effective Programs (REP) augmented with External Facilitation (EF)
  Interventions: Behavioral: External Facilitation
- REP + EF/IF (Experimental): Replicating Effective Programs (REP) augmented with External and Internal Facilitation (EF + IF)
  Interventions: Behavioral: External + Internal Facilitation

INTERVENTIONS:
Behavioral: External Facilitation — Non-responding sites randomized to receive external facilitation
  Arms: REP + EF
Behavioral: External + Internal Facilitation — Non-responding sites randomized to receive both internal and external facilitation
  Arms: REP + EF/IF

SUMMARY:
The overarching goal of this study is to build the most cost-effective adaptive implementation intervention involving a site-level implementation intervention strategy: Replicating Effective Programs (REP), and the augmentation of REP using either External Facilitation or a combination of an External and Internal Facilitation to improve patient outcomes and the uptake of an evidence-based program for mood disorders (Life Goals-LG) in community settings.

DETAILED DESCRIPTION:
Despite the availability of psychosocial evidence-based practices (EBPs), quality and outcomes for persons with mental disorders remain suboptimal because of organizational barriers to implementation. Replicating Effective Programs (REP), a site-level implementation strategy applied to promote the use of psychosocial treatments in community-based practices, still resulted in less than half of sites actually sustaining the use of these treatments. Based on input from community partners and previous research, the study team subsequently enhanced REP to include Facilitation, a novel implementation strategy which addresses site-level organizational barriers to EBP adoption beyond REP's emphasis on fidelity. Two Facilitation roles were developed: External and Internal Facilitators. External Facilitators (EFs) reside outside the clinic, are supported by the study, and provide technical expertise to providers in adapting and using EBPs in routine practice. Internal Facilitators (IFs) are employed by the sites, have a direct reporting relationship to site leadership, and have the local knowledge to help providers implement EBPs. IFs also address site-specific organizational barriers that may not be observable at baseline or by EFs. The overarching goal of this study is to build the most cost-effective adaptive implementation intervention involving REP and the augmentation of the EF and IF roles to improve patient outcomes and the uptake of an EBP for mood disorders (Life Goals-LG) in community settings. The primary aim of this clustered randomized trial is to determine, among sites not initially responding to REP (i.e., limited LG uptake), the effect of adaptive implementation interventions in sites receiving External and Internal Facilitator (REP+EF/IF) versus External Facilitator alone (REP+EF) on improved patient-level outcomes, including mental health quality of life and decreased symptoms, as well as increased LG use among patients with mood disorders after 12 months. Secondary aims are to determine, among sites that continue to exhibit non-response after 12 months, the effect of continuing Facilitation on patient-level outcomes at 24 months, describe the implementation of EF and IF, and to conduct a cost-effectiveness analysis of REP+EF/IF compared to REP+EF over the 24-month period. A representative cohort of 80 community-based outpatient clinics (total 1,600 patients) from different U.S. regions (Michigan, Colorado, and Arkansas) will be included in this study. We will use a Sequential Multiple Assignment Randomized Trial (SMART) design to build the best adaptive implementation intervention. This groundbreaking study design will address three crucial implementation issues: First, IFs are costly for sites since they require additional administrative effort. Second, the extent to which an off-site EF alone versus the addition of an on-site IF can improve patient outcomes in community settings is unclear. Finally, among sites that continue to exhibit non-response after 12 months of Facilitation, the value of continuing the implementation strategy (i.e., delayed effect) has not been assessed, especially in smaller practices from more rural settings.

ELIGIBILITY:
Inclusion Criteria:

* Currently being seen at one of the clinics participating in this study
* Diagnosis of or treated for a mood disorder (bipolar disorder or depression)
* Ability to speak and read English and provide informed consent

Exclusion Criteria:

* No active substance intoxication
* No acute medical illness or dementia

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2014-08; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Kilbourne, PhD, MPH, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Colorado Access, Denver, Colorado
  - University of Michigan, Ann Arbor, Michigan

REFERENCES:
- [Derived] Eisman AB, Hutton DW, Prosser LA, Smith SN, Kilbourne AM. Cost-effectiveness of the Adaptive Implementation of Effective Programs Trial (ADEPT): approaches to adopting implementation strategies. Implement Sci. 2020 Dec 14;15(1):109. doi: 10.1186/s13012-020-01069-w. PMID 33317593
- [Derived] Smith SN, Almirall D, Prenovost K, Liebrecht C, Kyle J, Eisenberg D, Bauer MS, Kilbourne AM. Change in Patient Outcomes After Augmenting a Low-level Implementation Strategy in Community Practices That Are Slow to Adopt a Collaborative Chronic Care Model: A Cluster Randomized Implementation Trial. Med Care. 2019 Jul;57(7):503-511. doi: 10.1097/MLR.0000000000001138. PMID 31135692
- [Derived] Kilbourne AM, Almirall D, Eisenberg D, Waxmonsky J, Goodrich DE, Fortney JC, Kirchner JE, Solberg LI, Main D, Bauer MS, Kyle J, Murphy SA, Nord KM, Thomas MR. Protocol: Adaptive Implementation of Effective Programs Trial (ADEPT): cluster randomized SMART trial comparing a standard versus enhanced implementation strategy to improve outcomes of a mood disorders program. Implement Sci. 2014 Sep 30;9:132. doi: 10.1186/s13012-014-0132-x. PMID 25267385

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 383 participants were consented and enrolled to participate. Of those 383 participants, only 169 were randomized participants from a non-responsive site.
Period: Overall Study
Arm/Group | REP + EF | REP + EF/IF
Started | 77 | 92
Completed | 45 | 52
Not Completed | 32 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REP + EF | REP + EF/IF | Total
Number analyzed (Participants) | 77 | 92 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (11.14) | 43.0 (11.19) | 45.38 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 71 | 125
  Male | 23 | 21 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 61 | 73 | 134
  Not Available | 16 | 19 | 35
Region of Enrollment [Number; unit: participants]
  United States | 77 | 92 | 169
Mental Health Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Mental Health Quality of Life was measured using the 12-Item Short Form Survey (SF-12). The SF-12 has a scale range of 0-100 with higher values representing better outcomes.
  units on a scale | 39.75 (12.92) | 36.66 (13.10) | 38.08 (13.07)
Mood Disorder Symptoms (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — Mood disorder symptoms were measured using the Patient Health Questionnaire (9-question). The PHQ-9 has a scale range of 0-27 with lower values representing better outcomes.
  units on a scale | 11.45 (6.46) | 12.61 (6.94) | 12.08 (6.73)

OUTCOME MEASURES:

1. Primary Outcome: Health-related Quality of Life - Mental Health Component Score
Description: Mental Health Quality of Life was measured using the 12-Item Short Form Survey (SF-12). The SF-12 has a scale range of 0-100 with higher values representing better outcomes.
Time Frame: Change from Baseline in Quality of Life at 12-months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | REP + EF | REP + EF/IF
Number analyzed (Participants) | 45 | 52
score on a scale | 2.14 [-0.22 to 4.50] | -0.20 [-3.25 to 0.86]

2. Primary Outcome: Reduced Mood Disorder Symptoms
Description: Mood disorder symptoms were measured using the Patient Health Questionnaire (9-question). The PHQ-9 has a scale range of 0-27 with lower values representing better outcomes.
Time Frame: Change from Baseline in Mood Disorder Symptoms at 12-months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | REP + EF | REP + EF/IF
Number analyzed (Participants) | 45 | 52
score on a scale | -1.57 [-2.65 to -0.50] | -1.02 [-2.02 to -0.01]

3. Secondary Outcome: Health-related Quality of Life - Mental Health Component Score
Description: Health-related Quality of Life - Mental Health Component Score of the short form (SF)-12 survey
Time Frame: Change from Baseline in Quality of Life at 24-months
Population: No analysis was completed because the funder requested terminating the study due to low enrollment. No data was collected because the study was halted prematurely.
Arm/Group | REP + EF | REP + EF/IF
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Reduced Mood Disorder Symptoms
Time Frame: Change from Baseline in Mood Disorder Symptoms at 24-months
Population: as for outcome 3
Arm/Group | REP + EF | REP + EF/IF
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected over an 18-month period
Description: No adverse events were reported for this study
Arm/Group | REP + EF | REP + EF/IF
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/92
Other Adverse Events (participants affected / at risk) | 0/77 | 0/92

LIMITATIONS AND CAVEATS:
Number of patients referred for study was much lower than anticipated; many sites participating in the study (N=18) did not refer any patients and therefore are not included in patient-level outcomes analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT02151331/Prot_SAP_000.pdf